CLINICAL TRIAL: NCT00784953
Title: Real Life Effectiveness in Patients With Not Optimally Controlled Asthma: Symbicort SMART, or Other ICS/LABA With as Needed SABA
Brief Title: Real Life Effectiveness in Patients With Not Optimally Controlled Asthma
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-RTW-SYM-2008/1
Record Dates: First submitted 2008-11-03; First posted 2008-11-04 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Asthma
Keywords: Symbicort SMART; budesonide; formoterol; ICS/LABA; Asthma Control Questionnaire; Not optimally controlled asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Asthma patients who were partly controlled or uncontrolled, need to step up, or adjust dose of the controller medications to ICS/LABA

SUMMARY:
A non-interventional study to explore actual asthma control status in real-life environment and to observe the efficacy after stepped-up to Symbicort SMART or various identical regimens.

The study will be implemented by screening asthmatic patients from respiratory clinics to identify those not optimally controlled and required stepping up the controllers to initiate, or to titrate dose of, ICS/LABA including Symbicort.

ELIGIBILITY:
Inclusion Criteria:

* Asthma patient who was partly controlled or uncontrolled by previous controllers of ICS only, or low dose ICS plus either LABA, leukotriene modifier or theophylline; or ICS- naïve with severe and persist symptom based on physician's judgment
* According to GINA guideline, who need to step up the controller medications, and ICS/LABA to be prescribed based on physician's discretion

Exclusion Criteria:

* Patients aged not within limitation refer to label information of various product prescribed
* Patients who have taken oral corticosteroids within 4 weeks prior to enrollment
* Patients with contraindications to prescribed medication

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Medical center
Sampling Method: Probability Sample
Enrollment: 842 (Actual)
Dates: Start 2008-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Change in ACQ score from baseline to the mean of all available data from the follow up visits | wk 4±1; wk 12~16

SECONDARY OUTCOMES:
Change in the individual asthma control status & pulmonary function from enrollment | wk 4±1; wk 12~16
Dose/usage of ICS/LABA and relievers & Patient compliance | wk 4±1; wk 12~16
Medical resource utilization | wk 4±1; wk 12~16; 6 month; 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Robin Meng, MD, PhD, Study Director — AstraZeneca Taiwan; Jia-Horng Wang, MD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (6):
- Taiwan (6):
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, Keelung
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei

REFERENCES:
- [Derived] Cheng SL, Ho ML, Lai YF, Wang HC, Hsu JY, Liu SF, Huang MS, Lee CH, Lin CH, Hang LW, Liu YC, Yang KY, Wang JH. Budesonide/Formoterol Anti-Inflammatory Reliever and Maintenance or Fluticasone Propionate/Salmeterol Plus As-Needed, Short-Acting beta2 Agonist: Real-World Effectiveness in pAtients without Optimally Controlled asThma (REACT) Study. Drug Des Devel Ther. 2020 Dec 8;14:5441-5450. doi: 10.2147/DDDT.S266177. eCollection 2020. PMID 33324041
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1082&filename=CSR-NIS-RTW-SYM-2008-1.pdf